CLINICAL TRIAL: NCT02264132
Title: A Multiple Dose Study of Pramipexole With Increasing Doses (0.375 mg to 1.5 mg q.d.) of Oral Extended Release (ER) Tablet in Two-way Cross-over Comparison of 0.375 mg ER Tablet q.d. Versus 0.125 mg Immediate Release (IR) Tablet t.i.d. and 1.5 mg ER Tablet q.d. Versus 0.5 mg IR Tablet t.i.d. in Japanese Healthy Male Volunteers
Brief Title: Increasing Dose Study of Pramipexole in Two-way Cross-over Comparison of ER Tablet Versus IR Tablet in Japanese Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 248.607
Record Dates: First submitted 2014-10-14; First posted 2014-10-15 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Healthy

ARMS (2):
- Pramipexole ER tablet versus Pramipexole IR tablet (Experimental)
  Interventions: Drug: Pramipexole ER tablet; Drug: Pramipexole IR tablet
- Pramipexole IR tablet versus Pramipexole ER tablet (Experimental)
  Interventions: Drug: Pramipexole ER tablet; Drug: Pramipexole IR tablet

INTERVENTIONS:
Drug: Pramipexole ER tablet
Drug: Pramipexole IR tablet

SUMMARY:
The objectives of this study were to investigate relative BA at steady state and to investigate dose proportionality of pharmacokinetic parameters

Relative BA at steady state:

* Pramipexole 0.375 mg ER tablet q.d. versus pramipexole 0.125 mg IR tablet t.i.d.
* Pramipexole 1.5 mg ER tablet q.d. versus pramipexole 0.5 mg IR tablet t.i.d.

Dose proportionality of pharmacokinetic parameters:

· Pramipexole ER dosages from 0.375 to 1.5 mg q.d.

ELIGIBILITY:
Inclusion Criteria:

* All subjects participating in the study are healthy male volunteers
* Age between 20 and 40 years
* Body mass index (BMI) between 17.6 and 26.4 kg/m2
* All volunteers must give written informed consent before screening to participate in this study and before first drug administration on Day 1 at Visit 2

Exclusion Criteria:

* Any findings of the medical examination (including blood pressure, pulse rate, ECG, and laboratory test parameters) of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy), psychiatric disorders or neurological disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (>24 hours) within at least one month or less than ten half-lives of the respective drug before the administration of investigational products
* Use of any drugs which might influence the results of the trial within 7 days before the start of drug administration in the study or during the study period
* Participation in another trial with an investigational drug (within 4 months before the start of drug administration)
* Smoker (>10 cigarettes or >3 cigars or >3 pipes/day and who cannot refrain from smoking at the trial site)
* Alcohol abuse (>40 g/day)
* Drug abuse
* Blood donation (≥100 mL within 4 weeks before drug administration or during the trial)
* Excessive physical activities from 7 days before the start of drug administration to the end of this study
* Any positive results in hepatitis B surface antigen (HBsAg), anti hepatitis B core (HBc) antibodies, anti hepatitis C virus (HCV) antibodies and human immunodeficiency virus (HIV) test

The following exclusion criteria are of special interest for this study:

* Hypersensitivity to pramipexole or other dopamine agonists
* Supine blood pressure at screening of systolic <110 mmHg and diastolic <60 mmHg

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2006-09; Primary Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
AUCτ,ss=AUC0-24,ss for ER (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ=24 hours) | up to day 5
AUC0-24,ss for IR (area under the concentration-time curve of the analyte in plasma over the time interval 0 to 24 hours at steady state) (This parameter was calculated as 3 times of AUC0-8,ss.) | up to 24 hours after drug administration

SECONDARY OUTCOMES:
Ae0-24,ss (amount of analyte that is eliminated in urine from 0 to 24 hours at steady state) | up to 24 hours after drug administration
  Relative BA
AUCτ,ss=AUC0-24,ss for ER (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ=24 hours) | up to 24 hours after drug administration
  Dose proportionality (only for ER)
Cmax,ss (maximum measured concentration of the analyte in plasma at steady state) | up to day 5
  Dose proportionality (only for ER)
Ae0-24,ss (amount of analyte that is eliminated in urine from 0 to 24 hours at steady state) | up to 24 hours after drug administration
  Dose proportionality (only for ER)
AUCτ,ss=AUC0-24,ss for ER (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ=24 hours) | up to 24 hours after drug administration
AUC0-24,ss for IR (area under the concentration-time curve of the analyte in plasma over the time interval 0 to 24 hours at steady state) (This parameter was calculated as 3 times of AUC0-8,ss.) | up to 24 hours after drug administration
Cmax,ss (maximum measured concentration of the analyte in plasma at steady state) | up to day 5
Cmin,ss (minimum measured concentration of the analyte in plasma at steady state) | up to day 5
PTF (peak-trough fluctuation) | up to day 5
tmax,ss (time from last dosing to the maximum concentration of the analyte in plasma at steady state) | up to day 5
Cpre,ss (predose concentration of the analyte in plasma at steady state immediately before administration of the next dose) | up to day 5
Cavg (average concentration of the analyte in plasma at steady state) | up to day 5
t1/2,ss (terminal half-life of the analyte in plasma at steady state) | up to day 5
CL/F,ss (apparent clearance of the analyte in plasma at steady state after | up to day 5
CLR,ss (renal clearance of the analyte at steady state determined over the dosing interval τ) | up to day 5
Vz/F,ss (apparent volume of distribution during the terminal phase λz at steady state following oral administration) | up to day 5
Ae0-24,ss (amount of analyte that is eliminated in urine from 0 to 24 hours at steady state) | up to 24 hours after drug administration
Ae0-8,ss for IR (amount of analyte that is eliminated in urine from 0 to 8 hours at steady state) | up to 8 hours after drug administration
AUC0-8,ss for IR (area under the concentration-time curve of the analyte in plasma over the time interval 0 to 8 hours at steady state) | up to 8 hours after drug administration
Number of subjects with adverse events | up to 7 days after last drug administration
Assessment of tolerability by investigator on a 4-point scale | Day 5